CLINICAL TRIAL: NCT02046733
Title: A Randomised Open-label Phase II Trial of Consolidation With Nivolumab and Ipilimumab in Limited-stage SCLC After Chemo-radiotherapy
Brief Title: Small Cell Lung Carcinoma Trial With Nivolumab and IpiliMUmab in LImited Disease
Acronym: STIMULI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Intergroupe Francophone de Cancerologie Thoracique (Other); Ludwig Center for Cancer Research of Lausanne (Other); Frontier Science Foundation, Hellas (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP/IFCT 4-12; 2013-002609-78 (EudraCT Number); CA184-310 (Other: Bristol-Myers Squibb); SNCTP000000166 (Registry Identifier: Swiss National Clinical Trials Portal (SNCTP))
Record Dates: First submitted 2014-01-17; First posted 2014-01-28 (Estimated); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-09

CONDITIONS: Limited Stage Small Cell Lung Cancer; Small Cell Lung Cancer
Keywords: SCLC; CTLA-4
MeSH Terms: conditions — Small Cell Lung Carcinoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nivolumab + Ipilimumab (Experimental): - Induction: Nivolumab at a dose of 1 mg/kg i.v. followed (on the same day) by Ipilimumab at a dose of 3 mg/kg i.v. once every 3 weeks, 4 cycles
  - Maintenance: Nivolumab 240 mg i.v. once every 2 weeks, for a maximum of 12 months from start of maintenance
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Observation (No Intervention): no further treatment; tumour assessment, follow-up documentation and collection of biological material will be done according to the same schedule as Arm 1.

INTERVENTIONS:
Drug: Ipilimumab — Induction phase: i.v. 3 mg/kg, once every 3 weeks × 4 cycles, to start within 6-8 weeks (42-56 days) from start of chemotherapy cycle 4, and not more than 2 weeks (14 days) after the date of randomisation)
  Other Names: Yervoy
  Arms: Nivolumab + Ipilimumab
Drug: Nivolumab — Induction phase: Nivolumab i.v. 1 mg/kg, once every 3 weeks × 4 cycles, to start within 6-8 weeks (42-56 days) from start of chemotherapy cycle 4, and not more than 2 weeks (14 days) after the date of randomisation) Maintenance Phase: Nivolumab 240 mg i.v once every 2 weeks for a maximum of 12 months from start of maintenance (the first dose of maintenance nivolumab will be administered 3 weeks after the last IMP doses of induction Phase).
  Other Names: Opdivo
  Arms: Nivolumab + Ipilimumab

SUMMARY:
Despite the fact that the majority of the patients with limited disease SCLC will respond very well to the standard treatment, a great proportion will relapse within 12 - 24 months.

Several studies in patients with lung cancer suggested a possible favourable association between the increased presence of immunologically active cells in the tumour and survival. Nivolumab and ipilimumab are proteins, which help your immune system to attack and destroy cancer cells by your immune cells. Early clinical trials with nivolumab and ipilimumab have shown activity in a broad range of cancers, including SCLC.

The aim of the current study is to investigate the efficacy (how well the treatment works) and tolerability (how severe the side effects are) of the standard treatment (chemotherapy and radiotherapy) alone, compared with the standard treatment followed by nivolumab and ipilimumab in patients with limited SCLC.

DETAILED DESCRIPTION:
At the time of diagnosis, 30% of patients with small cell lung carcinoma (SCLC) will have limited stage disease, now called stage I-IIIB (IASLC). The outcome of limited disease SCLC is still poor, with a median survival of 16 to 24 months with current forms of treatment and only 15-25% long term survivors.

Combining chemotherapy and thoracic radiotherapy is the standard treatment approach in limited-stage SCLC with a combination of platinum compounds (cis- or carboplatin) and etoposide and cisplatin (PE) as the backbone regimen. Concurrent chemo-radiotherapy is superior to sequential treatment and early thoracic irradiation starting with first or second cycle of chemotherapy appears beneficial. Hyperfractionated accelerated radiotherapy has been shown to be more efficacious than radiotherapy given in a long overall treatment time. However, availability and routine-use of hyperfractionated radiotherapy remains a matter of debate. Therefore, in this trial, both radiotherapy schedules of accelerated twice-daily administration or once-daily radiotherapy are accepted. The choice of schedule is a stratification factor for randomisation.

The adaptive immune response is triggered via effector T-cells, antigen-presenting cells (APCs) and co-stimulatory signals mediated by T cell receptors such as CD28. The interplay of these signals results in the activation and clonal proliferation of T cells.

T-cell proliferation is tightly regulated in order to avoid autoimmunity. The balance between co-stimulatory signals mediated by CD28 and co-inhibitory signals via so called immune checkpoint receptors is crucial for the maintenance of self-tolerance and to protect tissues from damage during normal immune response. After activation, T-cells express the immune checkpoint receptors cytotoxic T-lymphocyte antigen-4 (CTLA-4) and programmed cell death protein 1 (PD-1).

CTLA-4- and PD-1 expressing T-cells play a critical role in maintaining self-tolerance but are also responsible for non-responsiveness to tumour antigens. Cancer cells escape from im-mune surveillance by expressing immune checkpoint receptors. The goal of immune check-point inhibitor therapies is not to activate the immune system to attack particular targets on tumour cells, but rather to remove inhibitory pathways that block effective antitumour T cell responses.

Ipilimumab is a monoclonal antibody that binds to CTLA-4 and inhibits the interactions with the ligands B7.1 and B7.2, Nivolumab is a monoclonal antibody that targets PD-1. Engagement of PD-1 by its natural ligands, PD-L1 and PD-L2, results in an inhibition of T cell proliferation, survival and cyto-kine secretion. Nivolumab abrogates this interaction between PD-1 and its ligands.

The two antibodies, nivolumab and ipilimumab, do not only target different immune cell receptors, they also regulate distinct inhibitory pathways and have therefore non-overlapping mechanisms of action. Anti-CTLA-4 therapies seem to drive T-cells into tumours, resulting in an increased number of intratumour T-cells and a concomitant increase in IFN-y. This in turn can induce the expression of PD-L1 in the tumour microenvironment, with subsequent inhibition of antitumour T-cell responses, but may also increase the chance of benefit from anti-PD-1 and anti-PD-L1 therapies. A combination treatment with anti-CTLA-4 (e.g. ipili-mumab) plus anti PD-1 (e.g. nivolumab) or anti-PD-L1 antibodies should enable the creation of an immunogenic tumour microenvironment with subsequent clinical benefit for patients.

Nivolumab monotherapy has been approved for the treatment of advanced melanoma (FDA, EMA, and Japan) and previously treated squamous NSCLC (FDA, positive CHMP opin-ion). Nivolumab and ipilimumab improved PFS compared to nivolumab or ipilimumab alone in a study in melanoma (CA209067).

In a randomised open-label phase I/II trial (CheckMate 032), evaluating nivolumab with or without ipilimumab in pretreated SCLC patients with progressive disease and sensitive or refractory to platinum based chemotherapy, based on an interim analysis a response rate of 33% and disease stabilisation in 22% was observed for the combination of nivolumab and ipilimumab compared to 18% response rate and 20% stable disease with nivolumab mono-therapy.

Both, nivolumab monotherapy and nivolumab plus ipilimumab combination treatment were tolerable for the treatment of SCLC, and no new safety profile was identified compared to the profile of nivolumab with or without ipilimumab in other anti-cancer therapies.

Nivolumab plus ipilimumab will be administered as a consolidation treatment after comple-tion of a standard treatment including chemo-radiotherapy and prophylactic cranial irradia-tion (PCI).

ELIGIBILITY:
Inclusion Criteria for enrolment:

* Histologically or cytologically confirmed small cell lung carcinoma.
* Untreated limited-stage disease (with the exception of one cycle of chemotherapy given prior to enrolment) as defined by stage I-IIIB based on 7th TNM classification (IASLC classification for SCLC proposal). M0 proven by whole body FDG-PET CT including a contrast-enhanced CT of thorax and upper abdomen (incl. liver, kidney, adrenals); OR contrast-enhanced CT of thorax and upper abdomen (incl. liver, kidney, adrenals) and bone scan; AND brain MRI (or contrast enhanced CT of the brain) within 28 days before start of chemotherapy.
* Age ≥ 18 years.
* ECOG performance status 0-1.
* Adequate haematological function: haemoglobin > 9 g/dL, neutrophils count >1.5×109/L, platelet count > 100 × 109/L.
* Adequate liver function: total bilirubin < 2.5 × ULN, ALT and/or AST < 2.5 × ULN, alkaline phosphatase < 5 ULN.
* Adequate renal function: Calculated creatinine clearance ≥ 30 mL/min (Cockroft-Gault).
* Pulmonary function FEV1 of 1.0L or > 40% predicted value and DLCO > 40% predicted value.
* Patient capable of proper therapeutic compliance, and accessible for correct follow-up.
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before beginning of chemotherapy.
* All sexually active men and women of childbearing potential must use an effective contraceptive method (two barrier methods or a barrier method plus a hormonal method) during the study treatment and for a period of at least 12 months following the last administration of trial drugs.
* Measurable or evaluable disease (according to RECIST 1.1 criteria). Not eligible: patients with only one measurable or evaluable tumour lesion which was resected or irradiated prior to enrolment.
* Written Informed Consent (IC) must be signed and dated by the patient and the investigator prior to any trial-related intervention for a) Chemo-radiotherapy treatment and PCI, and subsequent randomisation, including mandatory biological samples b) Optional biological material collection, long-term storage and future use of biological material for translational research.

Exclusion Criteria for enrolment:

* Patient with mixed small-cell and non-small-cell histologic features.
* Patient with pleural or pericardial effusions proven to be malignant.
* Patients who have had in the past 5 years any previous or concomitant malignancy EXCEPT adequately treated basal or squamous cell carcinoma of the skin, in situ carcinoma of the cervix or bladder, in situ ductal carcinoma of the breast (if no RT was involved).
* Patients with other serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical processes that could affect the patient's capacity to participate in the study.
* Ongoing clinically serious infections requiring systemic antibiotic or antiviral, antimicrobial, antifungal therapy.
* Known or suspected hypersensitivity to nivolumab or ipilimumab or any of their excipients.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Documented history of severe autoimmune or immune mediated symptomatic disease that required prolonged (more than 2 months) systemic immunosuppressive (e.g. steroids) treatment, such as but not limited to ulcerative colitis and Crohn´s disease, rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, or autoimmune vasculitis (eg, Wegener's granulomatosis).
* Subjects with an autoimmune paraneoplastic syndrome requiring concurrent immunosuppressive treatment.
* Interstitial lung disease or pulmonary fibrosis.
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.
* Patients with any concurrent anticancer systemic therapy (except for chemotherapy cycle 1).
* HIV, active Hepatitis B or Hepatitis C infection.
* Previous radiotherapy to the thorax (prior to inclusion), including RT for breast cancer.
* Planned radiotherapy to lung of mean dose > 20 Gy or V20 > 35 %.
* Patients who received treatment with an investigational drug agent during the 3 weeks before enrolment in the study.
* Prior chemotherapy or radiotherapy for SCLC. Exception: one cycle of chemotherapy (as specified to section 10.2 of the protocol) may be administered prior to enrolment.

Inclusion Criteria for randomisation:

* Chemo-radiotherapy completed per protocol: 4 cycles of chemotherapy, ≥85% of PTV of thoracic radiotherapy, as well as completed, mandatory PCI.
* Non-PD after chemo-radiotherapy and PCI.
* ECOG performance status 0-2.
* Recovery of all adverse events to a grade ≤1, except for fatigue, appetite, oesophagitis and renal impairment (where ≤2 is allowed) and alopecia (any grade).
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before randomisation.

Exclusion criteria for randomisation:

* Less than 4 cycles of chemotherapy administered, less than 85% PTV of thoracic radiotherapy delivered, or PCI not completed.
* Progressive disease after chemo-radiotherapy and PCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2022-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange Peters, MD PhD, Study Chair — European Thoracic Oncology Platform (ETOP); Dirk De Ruysscher, MD PhD, Study Chair — Maastro Clinic, Maastricht, The Netherlands
Locations (61):
- Australia (10):
  - Bendigo Hospital, Bendigo
  - Coffs Harbour Health Campus, Coffs Harbour
  - Royal Brisbane and Women's Hospital (QLD), Herston
  - Royal Hobart Hospital, Hobart
  - NNSWLHD - The Tweed Hospital, Lismore
  - Austin Hospital, Melbourne
  - Riverina Cancer Centre, Mount Kuring-Gai
  - Port Macquarie Base Hospital, Port Macquarie
  - Epworth HealthCare - Richmond, Richmond
  - Princess Alexandra Hospital, Woolloongabba
- University Hospital Gasthuisberg, KU Leuven, Leuven, Belgium
- France (26):
  - Avignon - Institut Sainte-Catherine, Avignon
  - Caen - Centre François Baclesse, Caen
  - CHU, Caen
  - Percy/Armées, Clamart
  - Clermont-Ferrand, Clermont-Ferrand
  - Créteil - CHI, Créteil
  - CHU, Grenoble
  - Centre Hospitalier Général, Le Mans
  - Hôpital Louis Pradel, Lyon
  - Lyon - Sud, Lyon
  - AP-HM, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CH, Mulhouse
  - CRLCC, Nantes
  - Nice - CRLCC, Nice
  - Orléans - CH, Orléans
  - Paris - Bichat, Paris
  - Paris - Saint-Louis, Paris
  - Paris - Tenon, Paris
  - CHU, Rennes
  - Nouvel Hôpital Civil, Strasbourg
  - Suresnes, Suresnes
  - CHI, Toulon
  - CHU, Toulouse
  - CHU, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Klinikum Esslingen, Esslingen am Neckar
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Klinikum München-Bogenhausen, München
  - Thoracic Oncology Centre Munich, München
  - Pius-Hospital Oldenburg, Oldenburg
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitätsklinikum Tübingen, Tübingen
- Netherlands (2):
  - VUMC, Amsterdam
  - Maastro Clinic, Maastricht
- Spain (10):
  - Hospital General Universitario Alicante, Alicante
  - Hospital Universitario Cruces, Barakaldo
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Clinico San Carlos, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital Universitario Fundacion Jimenez Díaz, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
  - Hospital Virgen De La Salud, Toledo
  - Hospital Clínico Universitario De Valencia, Valencia
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - University Hospital Zürich, Zurich
- United Kingdom (3):
  - St James' University Hospital, Leeds
  - Royal Marsden, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lynch TJ, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Neal J, Lu H, Cuillerot JM, Reck M. Ipilimumab in combination with paclitaxel and carboplatin as first-line treatment in stage IIIB/IV non-small-cell lung cancer: results from a randomized, double-blind, multicenter phase II study. J Clin Oncol. 2012 Jun 10;30(17):2046-54. doi: 10.1200/JCO.2011.38.4032. Epub 2012 Apr 30. PMID 22547592
- [Background] Reck M, Bondarenko I, Luft A, Serwatowski P, Barlesi F, Chacko R, Sebastian M, Lu H, Cuillerot JM, Lynch TJ. Ipilimumab in combination with paclitaxel and carboplatin as first-line therapy in extensive-disease-small-cell lung cancer: results from a randomized, double-blind, multicenter phase 2 trial. Ann Oncol. 2013 Jan;24(1):75-83. doi: 10.1093/annonc/mds213. Epub 2012 Aug 2. PMID 22858559
- [Background] Margolin K, Ernstoff MS, Hamid O, Lawrence D, McDermott D, Puzanov I, Wolchok JD, Clark JI, Sznol M, Logan TF, Richards J, Michener T, Balogh A, Heller KN, Hodi FS. Ipilimumab in patients with melanoma and brain metastases: an open-label, phase 2 trial. Lancet Oncol. 2012 May;13(5):459-65. doi: 10.1016/S1470-2045(12)70090-6. Epub 2012 Mar 27. PMID 22456429
- See also: Sponsor — http://www.etop-eu.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From December 2015 to April 2019, a total of 222 patients were enrolled to the chemotherapy phase under protocol AM1 coming from 52 centers of 8 countries (France, Spain, Germany, Netherlands, Switzerland, United Kingdom, Belgium, and Australia). Overall, 153 patients were randomized under AM1 and constitute the ITT cohort of the efficacy analysis (145 of those were enrolled under AM1 and 8 were initially enrolled under the original protocol).
Groups:
- Observation: no further treatment; tumour assessment, follow-up documentation and collection of biological material will be done according to the same schedule as the experimental arm (nivolumab+ipilimumab).
- Nivolumab + Ipilimumab: * Induction phase to start within 6-8 weeks (42-56 days) after the start of chemotherapy cycle 4, and not more than 2 weeks (14 days) after the date of randomisation): Nivolumab at a dose of 1 mg/kg i.v. over a period of 30 minutes followed (on the same day) by Ipilimumab at a dose of 3 mg/kg i.v. over a period of 90 minutes once every 3 weeks (+/- 3 days, without dosing delay), for 4 cycles.
  * Maintenance phase (to start 3 weeks (21 days) after the last IMP dose of induction phase): Nivolumab 240 mg i.v. over a period of 30 minutes, once every 2 weeks (+/- 2 days, without dosing delay), for a maximum of 12 months from the start of maintenance phase.
Period: Overall Study
Arm/Group | Observation | Nivolumab + Ipilimumab
Started | 75 | 78
Completed | 69 | 78
Not Completed | 6 | 0
Not completed — never initiated 'treatment visits' | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation | Nivolumab + Ipilimumab | Total
Number analyzed (Participants) | 75 | 78 | 153
Age, Continuous [Median (Full Range); unit: years] — Age at enrolment
  years | 61.9 [38.6 to 77.3] | 61.1 [37.7 to 83.2] | 61.5 [37.7 to 83.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 28 | 61
  Male | 42 | 50 | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 7 | 7 | 14
  Belgium | 4 | 3 | 7
  United Kingdom | 1 | 3 | 4
  France | 24 | 31 | 55
  Australia | 2 | 3 | 5
  Switzerland | 5 | 4 | 9
  Germany | 9 | 7 | 16
  Spain | 23 | 20 | 43
Smoking history [Count of Participants; unit: Participants]
  Current | 25 | 27 | 52
  Former (≥ 100 cigarettes in the past during the whole life) | 49 | 51 | 100
  Never (0-99 cigarettes during the whole life) | 1 | 0 | 1
ECOG performance status (at randomization) [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction, 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work, 2: Ambulatory and capable of all self-care but unable to carry out any work activities; up and about more than 50% of waking hours, 3: Capable of only limited self-care; confined to bed or chair more than 50% of waking hours, 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair, 5: Dead
  Participants
    0 | 23 | 25 | 48
    1 | 51 | 50 | 101
    2 | 1 | 3 | 4
Stage [Count of Participants; unit: Participants] — Clinical stage is based on the 7th TNM classification (IASLC classification for SCLC proposal), which is the most widely used cancer staging system.
  Stage I: cancer has not grown deeply into nearby tissues and it also has not spread to the lymph nodes or other parts of the body (early-stage cancer).
  Stage II and III. In these 2 stages, cancers have grown more deeply into nearby tissue. They may have also spread to lymph nodes but not to other parts of the body.
  Stage IV. cancer has spread to other organs or parts of the body (advanced or metastatic cancer).
  Participants
    IA | 2 | 0 | 2
    IB | 1 | 2 | 3
    IIA | 5 | 3 | 8
    IIB | 2 | 6 | 8
    IIIA | 27 | 26 | 53
    IIIB | 36 | 40 | 76
    Missing | 2 | 1 | 3
Response to chemo-radiotherapy (before randomization) [Count of Participants; unit: Participants] — Response to chemo-radiotherapy treatment was assessed by RECIST1.1 criteria and done by the local radiologist; Complete Response(CR): Disappearance of all target lesions, Partial Response(PR): >=30% decrease in the sum of diameters of target lesions (reference the baseline sum of diameters, Progression(PD): At least a 20% increase in the sum of diameters of target lesions (reference the smallest sum recorded on the trial. Stable Disease(SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (reference the smallest sum of diameters recorded on the trial.
  Participants
    Complete response | 11 | 9 | 20
    Partial response | 60 | 65 | 125
    Stable disease | 3 | 4 | 7
    Not evaluable | 1 | 0 | 1
Number of radiotherapy fractions pre day [Count of Participants; unit: Participants]
  1 | 49 | 48 | 97
  2 | 26 | 30 | 56
PET-CT [Count of Participants; unit: Participants]
  Done | 26 | 25 | 51
  Not done | 49 | 53 | 102

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Defined as the time from the date of randomization until documented progression or death, if progression is not documented. Censoring for PFS occurs at the last tumor assessment.
  Assessment of Progressive Disease (PD) based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1):
  Target lesions: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on the study (this includes the baseline sum if that is the smallest on the study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Non-target lesions: Unequivocal progression of existing non-target lesions. To achieve 'unequivocal progression', there must be an overall level of substantial worsening in non-target disease such that, even in presence of SD or PR in target disease, the overall tumor burden has increased sufficiently.
  The appearance of one or more new lesions is also considered as progression.
Time Frame: From the date of randomization until documented progression (PD) according to RECIST v1.1 or death from any cause (whichever occurred first), up to 4.5 years.
Population: Intention-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Observation | Nivolumab + Ipilimumab
Number analyzed (Participants) | 75 | 78
months | 14.5 [8.2 to NA] — The upper 95% confidence limit for the median PFS time is not estimable because the upper limit of the survival curve hasn't reached 50%. | 10.7 [7.0 to NA] — The upper 95% confidence limit for the median PFS time is not estimable because the upper limit of the survival curve hasn't reached 50%.

2. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from the date of randomisation until death from any cause. Censoring for OS occurs at the last follow-up date.
Time Frame: From the date of randomization until death from any cause, up to 5.5 years.
Population: Intention-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Observation | Nivolumab + Ipilimumab
Number analyzed (Participants) | 75 | 78
months | 32.1 [26.1 to NA] — The upper 95% confidence limit for the median OS time is not estimable because the upper limit of the survival curve hasn't reached 50%. | NA [24.1 to NA] — Median OS is not reached (i.e survival curve doesn't cross 50% because survival is greater than 50% at the last time point) and the upper 95% confidence limit for the median OS time is not estimable because the upper limit of the survival curve hasn't reached 50%.

3. Secondary Outcome: Objective Response (OR)
Description: Objective response is defined as the best overall response (complete or partial response) according to RECIST 1.1 criteria across all assessment time-points during the period from randomisation to termination of trial treatment. Of note, the determination of OR is restricted to patients who have not attained a CR during the chemo-radiotherapy phase.
  Complete Response (CR): Disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum of diameters, Progression (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum recorded on the trial. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm., Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters recorded on the trial.
Time Frame: From randomisation to termination of trial treatment, for a maximum of 12 months from start of maintenance phase.
Population: Include only patients who have not attained a CR during the chemoradiotherapy phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Observation | Nivolumab + Ipilimumab
Number analyzed (Participants) | 64 | 69
Participants
  Complete response | 8 | 6
  Partial response | 22 | 20
  Stable disease | 22 | 28
  Progressive disease | 10 | 9
  Non-evaluable | 2 | 6

4. Secondary Outcome: Time-to-treatment Failure (TTF)
Description: Defined as the time from the date of randomisation to discontinuation of treatment for any reason (including progression of disease, treatment toxicity, refusal, lost to follow-up, and death). Censoring for TTF occurs at the last follow-up date.
Time Frame: From the date of randomization to treatment failure for any reason, up to 4.5 years.
Population: Intention-to-treat (ITT) population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Observation | Nivolumab + Ipilimumab
Number analyzed (Participants) | 75 | 78
months | 14.5 [8.2 to 24.0] | 1.7 [1.2 to 2.5]

5. Secondary Outcome: Adverse Events
Description: Adverse events graded according to NCI CTCAE V4.0.
Time Frame: Adverse events were assessed from randomization to 100 days after the last dose of study treatment, up to 4.5 years.
Population: Safety population, i.e., all patients who have received at least one dose of study treatment in the experimental arm (nivolumab_ipilimumab) plus all patients randomised to observation arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Observation | Nivolumab + Ipilimumab
Number analyzed (Participants) | 75 | 78
Participants
  Experienced AE/SAE | 65 | 77
  Not experienced AE/SAE | 10 | 1

ADVERSE EVENTS:
Time Frame: Reported adverse events (AEs) were assessed from randomization to 100 days after the last dose of study treatment, up to 4.5 years. Only all-cause mortality was from randomization up to 5.5 years.
Arm/Group | Observation | Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 37/75 | 34/78
Serious Adverse Events (participants affected / at risk) | 12/75 | 48/78
Other Adverse Events (participants affected / at risk) | 62/75 | 72/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=75) | Nivolumab + Ipilimumab (N=78)
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Syndrome of inappropriate antidiuretic hormone secretion (SIADH) (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 3
Hypothyroidism (Endocrine disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 8
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Fever (General disorders) | 0 | 3
Flu like symptoms (General disorders) | 0 | 1
Gait disturbance (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 0 | 1
Bronchial infection (Infections and infestations) | 0 | 2
Viral meningitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 2 | 6
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 2
Facial nerve disorder (Nervous system disorders) | 0 | 3
Polyneuropathy (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observation (N=75) | Nivolumab + Ipilimumab (N=78)
Anemia (Blood and lymphatic system disorders) | 13 | 7
Hyperthyroidism (Endocrine disorders) | 0 | 19
Hypothyroidism (Endocrine disorders) | 0 | 12
Abdominal pain (Gastrointestinal disorders) | 1 | 7
Constipation (Gastrointestinal disorders) | 3 | 14
Diarrhea (Gastrointestinal disorders) | 6 | 14
Dry mouth (Gastrointestinal disorders) | 0 | 6
Dysphagia (Gastrointestinal disorders) | 2 | 4
Mucositis oral (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 6 | 18
Vomiting (Gastrointestinal disorders) | 5 | 20
Chills (General disorders) | 1 | 5
Fatigue (General disorders) | 21 | 38
Fever (General disorders) | 1 | 8
Pain (General disorders) | 9 | 9
Lung infection (Infections and infestations) | 2 | 4
Upper respiratory infection (Infections and infestations) | 2 | 4
Urinary tract infection (Infections and infestations) | 3 | 7
Alanine aminotransferase increased (Investigations) | 1 | 6
Aspartate aminotransferase increased (Investigations) | 1 | 5
Platelet count decreased (Investigations) | 5 | 4
Weight loss (Investigations) | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 12 | 23
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (Nervous system disorders) | 8 | 9
Headache (Nervous system disorders) | 2 | 11
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 7
Depression (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 20
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 19
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 10

LIMITATIONS AND CAVEATS:
Because of the low accrual rate, as well as additional internal strategic considerations unrelated to the scientific rational or trial design, Bristol-Myers Squibb (BMS) decided not to continue funding the STIMULI trial. Thus, the trial Steering Committee decided to close the accrual permanently as of April 30, 2019. The statistical design was modified and the primary endpoint of the trial was finally defined as only the PFS (previous: co-primary PFS and OS).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/33/NCT02046733/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT02046733/SAP_001.pdf